CLINICAL TRIAL: NCT03659500
Title: Clinical Outcomes and Costs of 4-Week Versus 6-Week Bloodwork for Patients on Hemodialysis
Status: Completed | Type: Observational
Sponsor: Samuel Silver (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Samuel Silver, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: HD Lab Frequency 1
Record Dates: First submitted 2018-08-29; First posted 2018-09-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Four-week routine bloodwork: Routine bloodwork every 4-weeks (CBC, electrolytes, iron studies, calcium, phosphate, PTH) from June 1, 2012 to March 23, 2014
  Interventions: Diagnostic Test: Four-week routine bloodwork
- Six-week routine bloodwork: Routine bloodwork every 6-weeks (CBC, electrolytes, iron studies, calcium, phosphate, PTH) from March 25, 2014 to December 31, 2015
  Interventions: Diagnostic Test: Six-week routine bloodwork

INTERVENTIONS:
Diagnostic Test: Four-week routine bloodwork — Routine hemodialysis bloodwork done every 4 weeks
  Groups: Four-week routine bloodwork
Diagnostic Test: Six-week routine bloodwork — Routine hemodialysis bloodwork done every 6 weeks
  Groups: Six-week routine bloodwork

SUMMARY:
The objective of this quality improvement study was to determine the effect of an institution-wide switch of routine bloodwork from four-week intervals to six-week intervals on the achievement of anemia and chronic kidney disease-mineral and bone disorder (CKD-MBD) targets for patients on chronic hemodialysis.

DETAILED DESCRIPTION:
Rationale & Objective: Routine bloodwork for patients on hemodialysis has both financial and opportunity costs, but there is little data on how the frequency of measurement affects patient outcomes. Our objective was to determine the effect of changing from routine bloodwork at four-week intervals to six-week intervals on the achievement of anemia and chronic kidney disease-mineral and bone disorder (CKD-MBD) targets.

Study Design: Retrospective interrupted time series from June 1, 2012 to December 31, 2015.

Setting & Participants: Tertiary hospital in Ontario, Canada, that provides hemodialysis to 350-400 adult patients.

Quality Improvement Activities: Institution-wide switch of routine bloodwork from four-week intervals to six-week intervals on March 24, 2014.

Outcomes: Proportion of patients who achieved recommended hemoglobin and phosphate targets. In a 252-day sub-analysis, we also calculated the cost-savings attributable to a change in laboratory testing frequency for hemoglobin, ferritin, iron saturation, calcium, and phosphate.

Analytical Approach: Statistical Process Control to analyze variation in the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all patients who received chronic hemodialysis at the Kingston Health Sciences Center regional hemodialysis program

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients on chronic hemodialysis at a regional hemodialysis program in Kingston, Ontario, Canada, from June 1, 2012 to December 31, 2015
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin target achievement | 650 days
  Proportion of patients who achieved hemoglobin (10-12 g/dl)
Phosphate target achievement | 650 days
  Proportion of patients who achieved phosphate (2.5-4.6 mg/dl)

SECONDARY OUTCOMES:
Use of erythropoietin | 650 days
  Proportion of patients on erythropoietin
Calcium target achievement | 650 days
  Proportion of patients with calcium (8.8-10.2 mg/dl)
PTH target achievement | 650 days
  Proportion of patients with PTH (94-462 pg/ml)
All-cause mortality | 650 days
  All-cause mortality

OTHER OUTCOMES:
Cost of laboratory tests | 650 days
  Direct costs (in CAD) of hemoglobin ($8.27), ferritin ($14.48), iron saturation ($17.58), serum calcium ($2.59), and serum phosphate ($2.59) based on the Ontario Schedule of Benefits for Laboratory Services

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Silver, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silver SA, Alaryni A, Alghamdi A, Digby G, Wald R, Iliescu E. Routine Laboratory Testing Every 4 Versus Every 6 Weeks for Patients on Maintenance Hemodialysis: A Quality Improvement Project. Am J Kidney Dis. 2019 Apr;73(4):496-503. doi: 10.1053/j.ajkd.2018.10.008. Epub 2018 Dec 28. PMID 30598347